CLINICAL TRIAL: NCT03086161
Title: Mood and Excess Weight Gain in Adolescent Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Colorado, Denver (Other); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-1505
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obesity; Adolescent Development; Pregnancy Related; Insulin Sensitivity; Interpersonal Relations; Stress
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Care providers delivering usual prenatal care are unaware of condition assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-as-usual (Active Comparator): Treatment-as-usual alone provided in the context of a multi-disciplinary teen pregnancy clinic providing wrap-around medical, nutrition, and social work care.
  Interventions: Behavioral: Treatment-as-usual
- Interpersonal Psychotherapy (Experimental): Treatment-as-usual plus a six-session interpersonal psychotherapy program delivered as individual sessions by a trained facilitator every 2-3 weeks throughout pregnancy.
  Interventions: Behavioral: Interpersonal Psychotherapy; Behavioral: Treatment-as-usual

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy — Six individual 1-hour sessions delivered over the course of pregnancy to address interpersonal problems areas that may lead to emotional eating, physical inactivity, and increased stress during pregnancy, which are drivers of excess weight gain in pregnancy
  Arms: Interpersonal Psychotherapy
Behavioral: Treatment-as-usual — Routine prenatal care as part of multidisciplinary adolescent pregnancy clinic, including medical (ob/gyn), nutrition, and social work

SUMMARY:
50-70% of adolescents gain too much weight during pregnancy, and this excess gain significantly increases their risk of high postpartum weight retention and long-term obesity. In this randomized controlled pilot study, the investigators are evaluating the feasibility and acceptability of a relatively brief interpersonal psychotherapy program for reducing excess gestational weight gain during adolescent pregnancy. Compared to treatment-as-usual prenatal care delivered in an adolescent maternity clinic, the investigators will estimate the added benefit of an interpersonal psychotherapy program's effectiveness for reducing excess gestational weight gain, improving maternal postpartum insulin sensitivity, and decreasing maternal and infant adiposity.

DETAILED DESCRIPTION:
Obesity and its negative health consequences such as type 2 diabetes and heart disease are major public health concerns. Pregnancy is an ideal opportunity to intervene with young women both to reduce their own likelihood of long-term obesity and to potentially lessen their offspring's obesity risk. Interventions to reduce excessive weight gain during adolescent pregnancy may be particularly important. 50-70% of adolescents gain too much weight during pregnancy, and this excess gain significantly increases their risk of high postpartum weight retention and long-term obesity. Depression and stress-which are common in adolescent pregnancy-also may play a role. Pregnant adolescent females, as well as non-pregnant females, who have more frequent feelings of depression or stress are more likely to gain weight too rapidly or to gain too much weight as they grow. In the current project, the investigators seek to develop a program to prevent excess weight gain that will be feasible to administer in the Colorado Adolescent Maternity Program (CAMP) at Children's Hospital Colorado, University of Colorado Denver, Anschutz Medical Campus, and, that will be acceptable to pregnant teens at-risk for gaining too much weight. After a screening assessment, adolescent females (13-19y) will be randomly assigned to participate in either a 6-session interpersonal psychotherapy (IPT) program + usual care or to CAMP usual care only. The IPT program will involve 6 1-hour meetings with a trained facilitator and focus on improving relationships, mood, stress, and eating in response to negative feelings. The investigators will assess participants midway through the program, immediately after the program, and again at a 3-month postpartum follow-up. The investigators will evaluate to what extent adolescent females attend the program, complete at-home practice assignments, and show changes in mood, stress, relationships, eating, and mindfulness before and after IPT participation compared to usual care only. The investigators also will estimate how program participation relates to weight gain during pregnancy and 3-month postpartum maternal weight retention, adiposity, and insulin sensitivity. The investigators also will study the adiposity of adolescents' 3-month-old infants.

ELIGIBILITY:
Inclusion Criteria:

* 13-19 years of age and the 3-6 month old infants of these adolescent mothers
* Female
* Pregnant, 12-18 weeks gestation
* Patient in the Colorado Adolescent Maternity Program (CAMP) clinic

Exclusion Criteria:

* Full-syndrome Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 psychiatric disorder that, in the opinion of the investigators, would impede study compliance and necessitate more intensive treatment (e.g., conduct disorder, schizophrenia, major depressive disorder with active suicidal ideation)
* Major renal, hepatic, endocrinologic (hyperthyroidism or Cushing syndrome), or pulmonary (other than mild asthma) disorder
* Medication affecting mood or body weight
* Major high-risk pregnancy complication (preeclampsia, gestational diabetes, hypertension, multiple gestation, placenta previa, membrane rupture, incompetent cervix)
* Pre-pregnancy BMI <5th percentile for age and sex

Ages: 3 Months to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | 5-year period
  Rate of recruitment
Acceptability | 6-9 months
  Program session attendance measured as percentage of total sessions (6) attended
Acceptability of program | 6-9 months
  Program acceptability ratings

SECONDARY OUTCOMES:
Depressive symptoms | 12 months (9 months of pregnancy plus 3 months postpartum)
  Depressive symptoms measured on the Center for Epidemiologic Studies Depression Scale
Perceived stress | 12 months (9 months of pregnancy plus 3 months postpartum)
  Perceived stress measured on the Perceived Stress Scale
Excess gestational weight gain | 9 months
  Weight gained from first-trimester screening to post-intervention assessment, just prior to delivery
Maternal postpartum insulin sensitivity | 12 months (9 months of pregnancy plus 3 months postpartum)
  Maternal postpartum insulin sensitivity
Maternal postpartum adiposity | 12 months (9 months of pregnancy plus 3 months postpartum)
  Maternal postpartum body fat percentage
Infant adiposity | Infants: 3 months
  Infant body fat percentage

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B Shomaker, PhD, Principal Investigator — Colorado State University
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shomaker LB, Gulley LD, Clark ELM, Hilkin AM, Pivarunas B, Tanofsky-Kraff M, Nadeau KJ, Barbour LA, Scott SM, Sheeder JL. Protocol for a pilot randomized controlled feasibility study of brief interpersonal psychotherapy for addressing social-emotional needs and preventing excess gestational weight gain in adolescents. Pilot Feasibility Stud. 2020 Mar 20;6:39. doi: 10.1186/s40814-020-00578-1. eCollection 2020. PMID 32206334